CLINICAL TRIAL: NCT05398003
Title: Evaluation of Multimodal Medullary Stimulation in Refractory Neck and Upper Limb Pain
Brief Title: Medullary Stimulation for the Treatment of Refractory Neck Pain (S2M)
Acronym: S2M
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RC21_0338
Record Dates: First submitted 2022-05-20; First posted 2022-05-31 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Pain, Intractable
Keywords: Medullary stimulation; refractory neck pain
MeSH Terms: conditions — Pain, Intractable; Neck Pain

STUDY DESIGN:
Intervention Model Description: Hierarchical sequential study with a fixed sequence of 3 successive hypotheses = tested with a 5% risk until one hypothesis is rejected. These three successive hypotheses are a non-inferiority test, followed by two superiority tests.
Masking Description: Patients will only know the stimulation modes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study population (Experimental): 12 patients with neck and upper limb pain who have failed multidisciplinary treatment and are candidates for cervical medullary stimulation will be included.
  Interventions: Device: Implantation of the WAVEWRITER ALPHA ™ device

INTERVENTIONS:
Device: Implantation of the WAVEWRITER ALPHA ™ device — The 12 patients will be implanted by the WAVEWRITER ALPHA ™ device. Then, the order of the three stimulation modes will be randomly selected and will be composed of 5 modalities:
  * tonic stimulation "LF": In tonic mode, the electrical stimulation of the sensory fibres of the posterior cords of the spinal cord induces local paresthesias
  * high frequency" stimulation (1000 Hz) "High Frequency".
  * stimulation in bursts (or "Burst")

SUMMARY:
Number of centres planned : 1 (CHU Nantes)

Design : Randomized, Prospective

Planning of the study :

* Total duration: 34 months
* Recruitment period: 24 months.
* Follow-up time per patients : 7-10 months

Expected number of cases : 12

Treatment, procedure, combination of procedures under consideration :

During the study, patients will be implanted with the WAVEWRITER ALPHA™ system with the objective of decreasing patient pain with a spinal cord stimulation mode.

There will be a random draw on the order of the stimulation program:

* the tonic stimulation "LF": In tonic mode, the electrical stimulation of the sensory fibers of the posterior cords of the spinal cord induces local paresthesias
* burst stimulation (or "burst")
* high frequency" stimulation (1000 Hz) "High frequency: HF".
* combined tonic + burst stimulation
* combined tonic + high frequency stimulation

ELIGIBILITY:
Inclusion criteria:

* Patients aged 18 to 85 years
* Patients with chronic neck and upper limb pain (according to HAS criteria for spinal cord stimulation)
* Patients must be able to give informed consent and must have signed an informed consent
* Affiliation to the health insurance
* A negative pregnancy test for women of childbearing potential
* Women of childbearing potential must use an appropriate contraceptive method(s) during the clinical trial

Non-inclusion criteria:

* Drug or alcohol abuse
* Any medical or psychological problem that may interfere with the proper conduct of the study protocol (e.g., cancer with limited life expectancy)
* Difficulty with follow-up
* Pregnant or breastfeeding women
* Women of childbearing potential who are not using contraception
* Adults under legal protection (guardianship, curatorship, "sauvegarde de justice") or deprived of liberty
* Exclusion period for another study
* Participation in another interventional study whose primary objective is based on pain.

Exclusion criteria:

- 7-day post-implantation test phase negative

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2026-09-23 (Estimated); Study Completion 2026-09-23 (Estimated)

PRIMARY OUTCOMES:
Evaluating the non-inferiority of pain reduction with the combined mode compared to the low frequency reference mode. | 6 Months
  Comparison of the average of the visual analogic scale (scale from 0 to 10 ; 10 being the worst outcome)score collected during the 7 days of stimulation by the Tonic+Burst mode to the average of the visual analogic scale score collected during the 7 days in tonic stimulation
Evaluating the overall satisfaction with the stimulation mode | 6 Months
  Daily collection of the patient's evaluation of his satisfaction on the remote control - the patient's logbook by a number of stars: 1* (one star) not satisfied and 5* (five stars) very satisfied
Evaluating the superioty of pain reduction with the combined mode compared to the low frequency reference mode. | 6 Months
  Comparison of the average visual analogic scale (scale from 0 to 10 ; 10 being the worst outcome) score of the 7 days of the Tonic+Burst mode compared to the average visual analogic scale scores collected in Tonic stimulation alone.

SECONDARY OUTCOMES:
Evaluating the non-inferiority of patient pain with the combined mode compared to the low frequency reference mode | 6 Months
  Comparison of the average of the visual analogic scale (scale from 0 to 10 ; 10 being the worst outcome) scores collected during the 7 days of stimulation by the combined Tonic+High Frequency mode to the average of the visual analogic scale scores collected during the 7 days of tonic stimulation.
Evaluating the non-inferiority of patient satisfaction with their overall comfort | 6 Months
  Daily collection of the patient's evaluation of his satisfaction on the patient's notebook by a number of stars: 1* (one star) not satisfied and 5* (five stars) very satisfied. During the 7 days of stimulation by Low frequency + High frequency.
Evaluating the superioty of pain reduction with the combined mode compared to the low frequency reference mode. | 6 Months
  Comparison of the average visual analogic scale (scale from 0 to 10 ; 10 being the worst outcome) score of the 7 days of the combined mode Tonic+ High Frequency compared to the average visual analogic scale scores collected in Tonic stimulation alone
Evaluating the non-inferiority of patient satisfaction with their overall comfort with the mode low frequency + burst vs Low frequency | 6 Months
  Daily collection of the patient's evaluation of his or her satisfaction on the patient logbook by a number of stars: 1* (one star) not satisfied and 5* (five stars) very satisfied.
Evaluating the non-inferiority of patient satisfaction with their overall comfort with the mode low frequency + high frequency vs Low frequency | 6 Months
  Daily collection of the patient's evaluation of his or her satisfaction on the patient logbook by a number of stars: 1* (one star) not satisfied and 5* (five stars) very satisfied.
Evaluating the superioty of pain reduction with the combined mode (low frequency + high frequency) compared to the tonic mode (low frequency) only | 6 Months
  Daily collection of the pain felt during the day (visual analogic scale (scale from 0 to 10 ; 10 being the worst outcome)) during the 7 consecutive days of stimulation of the same mode.
Evaluating the superioty of pain reduction with the combined mode (low frequency + Burst) compared to the tonic mode (low frequency) only | 6 Months
  Daily collection of the pain felt during the day (visual analogic scale (scale from 0 to 10 ; 10 being the worst outcome)) during the 7 consecutive days of stimulation of the same mode.
Evaluate the equality of the effectiveness of the new modes (Burst, high frequency, Tonic + Burst, Tonic + high frequency) compared to the tonic mode alone on the pain criteria | 6 Months
  Daily collection of the pain felt during the day (visual analogic scale (scale from 0 to 10 ; 10 being the worst outcome)) during the 7 consecutive days of stimulation of the same mode.
Evaluate the equality of the effectiveness of the new modes (Burst, high frequency, Tonic + Burst, Tonic + high frequency) compared to the tonic mode alone on the satisfaction | 6 Months
  Daily collection of the patient's evaluation of his or her satisfaction on the patient logbook by a number of stars: 1* (one star) not satisfied and 5* (five stars) very satisfied.
Comparison of the number of recharges of the device according to the stimulation modes | 6 Months
  Number of recharges of the remote control during the 7 days of stimulation.
Evaluating the change in the quality of life of patients at 1 month | 1 month
  Comparison of the evolution of quality of life from inclusion to 1 month with the Hospital Anxiety and Depression scale (scale from 0 to 3; 3 being the worst outcome)
Evaluating the change in the quality of life of patients at 1 month | 1 month
  Comparison of the evolution of quality of life from inclusion to 1 month with the EuroQol 5 Dimensions (scale from 0 to 100; 100 being the worst outcome)
Evaluating the change in the quality of life of patients at 3 months | 3 months
  Comparison of the evolution of quality of life from inclusion to 3 months with the Hospital Anxiety and Depression scale (scale from 0 to 3; 3 being the worst outcome)
Evaluating the change in the quality of life of patients at 3 months | 3 months
  Comparison of the evolution of quality of life from inclusion to 3 months with the EuroQol 5 Dimensions (scale from 0 to 100; 100 being the worst outcome)
Evaluating the change in the quality of life of patients at 6 months | 6 months
  Comparison of the evolution of quality of life from inclusion to 6 months with the Hospital Anxiety and Depression scale (scale from 0 to 3; 3 being the worst outcome)
Evaluating the change in the quality of life of patients at 6 months | 6 months
  Comparison of the evolution of quality of life from inclusion to 6 months with the EuroQol 5 Dimensions (scale from 0 to 100; 100 being the worst outcome)
Evaluating average daily analgesic consumption at inclusion. | 0 month
  Collection of the number and type of analgesic treatments per day for one week prior to the inclusion visit with the Medication Quantification Scale (scale from 0 to 36; 36 being the worst outcome) .
Evaluating average daily analgesic consumption at 1 month | 1 month
  Collection of the number and type of analgesic treatments per day for one week prior to the month 1 visit with the Medication Quantification Scale (scale from 0 to 36; 36 being the worst outcome) .
Evaluating average daily analgesic consumption at 3 months | 3 month
  Collection of the number and type of analgesic treatments per day for one week prior to the month 3 visit with the Medication Quantification Scale (scale from 0 to 36; 36 being the worst outcome) .
Evaluating average daily analgesic consumption at 6 months | 6 month
  Collection of the number and type of analgesic treatments per day for one week prior to the month 6 visit with the Medication Quantification Scale (scale from 0 to 36; 36 being the worst outcome) .

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No